CLINICAL TRIAL: NCT01005667
Title: Management of Labor Using the BirthTrack Computerized Labor Monitoring System
Brief Title: Study to Determine if Monitoring of Labor Shortens the Time to Delivery
Acronym: BirthTrack
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding for the company has resulted in termination of the study.
Sponsor: Barnev, Inc. (Industry)
Responsible Party: John Quigley, Barnev, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BBT1600
Record Dates: First submitted 2009-10-30; First posted 2009-11-02 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2009-10

CONDITIONS: Pregnancy
Keywords: Nulliparous women in spontaneous labor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BirthTrack Monitor (Experimental)
  Interventions: Device: BirthTrack
- Control - no BirthTrack Monitor (No Intervention)

INTERVENTIONS:
Device: BirthTrack — Measurement of cervical dilation and head station
  Other Names: Computerized Labor Monitoring System
  Arms: BirthTrack Monitor

SUMMARY:
The purpose of this study is to test the hypothesis that using the BirthTrack for management of labor shortens the time to delivery and thus improves both maternal and perinatal outcomes.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be ≥ 18 years old
* Nulliparous
* Singleton fetus in vertex presentation
* Gestational age 36-0/7 or more
* Reassuring fetal heart tracing

Exclusion Criteria:

* Any significant medical condition which in the Investigator's opinion may interfere with the patient's optimal participation in the study
* Low lying placenta (edge 3cm or less from cervix)
* Known or suspected fetal or maternal infection
* Maternal thrombocytopenia (platelet count <100,000)
* Maternal bleeding disorder
* Women with previous uterine surgery
* Known major fetal malformation
* Suspected fetal growth restriction (EFW<10th percentile)
* Subjects with significant psychiatric history
* Major maternal morbidity (e.g. major cardiac disease)
* Subjects with indication for immediate delivery
* Limit on cervical dilation (e.g., up to 7 cm.)
* Prolonged rupture of membranes (i.e., > 24 hours)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)

PRIMARY OUTCOMES:
Shortened time to vaginal delivery | Length of labor until delivery

CONTACTS AND LOCATIONS:
Overall Officials: Barak M Rosenn, MD, Principal Investigator — St. Luke's-Roosevelt Hospital Center; Dan Farine, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada